CLINICAL TRIAL: NCT02544230
Title: Efficacy of Granulocyte Transfusions for the Treatment of Severe Infections in Hematological Patients With Febrile Neutropenia
Brief Title: Granulocyte Transfusions in Hematological Patients With Febrile Neutropenia
Status: Completed | Type: Observational
Sponsor: Sorveglianza Epidemiologica Infezioni Fungine Emopatie Maligne (Other)
Responsible Party: Principal Investigator, LIVIO PAGANO, Professor, Sorveglianza Epidemiologica Infezioni Fungine Emopatie Maligne
Other Study IDs: GTX.01
Record Dates: First submitted 2015-09-04; First posted 2015-09-09 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Neutropenia; Fever; Bacterial Infection; Fungal Infection; Fever of Unknown Origin; Hematological Neoplasms; Sepsis
Keywords: granulocyte transfusions
MeSH Terms: conditions — Neutropenia; Fever; Bacterial Infections; Mycoses; Fever of Unknown Origin; Hematologic Neoplasms; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators retrospectively evaluated the efficacy of granulocyte transfusions as adjunctive treatment for severe infections in neutropenic fever unresponsive to antimicrobial therapy in hematological patients.

ELIGIBILITY:
Inclusion Criteria:

* fever;
* presence of absolute neutrophil count <0.5 x 10^9/L
* evidence of bacterial or fungal infections (including clinical signs of infection, positive cultures or biopsy, and radiological evidences)
* unresponsiveness to appropriate antimicrobial therapy for at least 48 hours

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with malignant emopatia who received granulocyte transfusions as adjunctive therapy in the treatment of severe infection, unresponsive to appropriate antimicrobial therapy, which was incurred during neutropenia.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2004-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Infection-related mortality | within 30 days after the last granulocyte transfusion
  deaths due to infection occurred within 30 days after the last granulocyte transfusion

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Sacred Heart, Rome, Italy

REFERENCES:
- [Background] Estcourt LJ, Stanworth S, Doree C, Blanco P, Hopewell S, Trivella M, Massey E. Granulocyte transfusions for preventing infections in people with neutropenia or neutrophil dysfunction. Cochrane Database Syst Rev. 2015 Jun 29;2015(6):CD005341. doi: 10.1002/14651858.CD005341.pub3. PMID 26118415
- [Background] Stanworth SJ, Massey E, Hyde C, Brunskill S, Lucas G, Navarrete C, Marks DI. Granulocyte transfusions for treating infections in patients with neutropenia or neutrophil dysfunction. Cochrane Database Syst Rev. 2005 Jul 20;(3):CD005339. doi: 10.1002/14651858.CD005339. PMID 16034970
- [Background] Strauss RG. Role of granulocyte/neutrophil transfusions for haematology/oncology patients in the modern era. Br J Haematol. 2012 Aug;158(3):299-306. doi: 10.1111/j.1365-2141.2012.09190.x. Epub 2012 Jun 19. PMID 22712550
- [Background] Dale DC, Price TH. Granulocyte transfusion therapy: a new era? Curr Opin Hematol. 2009 Jan;16(1):1-2. doi: 10.1097/MOH.0b013e32831d7953. No abstract available. PMID 19057197
- [Background] Lee JJ, Chung IJ, Park MR, Kook H, Hwang TJ, Ryang DW, Kim HJ. Clinical efficacy of granulocyte transfusion therapy in patients with neutropenia-related infections. Leukemia. 2001 Feb;15(2):203-7. doi: 10.1038/sj.leu.2402007. PMID 11236935
- [Background] Ofran Y, Avivi I, Oliven A, Oren I, Zuckerman T, Bonstein L, Rowe JM, Dann EJ. Granulocyte transfusions for neutropenic patients with life-threatening infections: a single centre experience in 47 patients, who received 348 granulocyte transfusions. Vox Sang. 2007 Nov;93(4):363-9. doi: 10.1111/j.1423-0410.2007.00971.x. PMID 18070282